CLINICAL TRIAL: NCT00534794
Title: A Single-Center, Masked, Randomized Study Comparing Two Marketed Ocular Anti-Allergy Medications in the Cat Room Model
Brief Title: Study of Two Marketed Ocular Anti-Allergy Medications in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 031-408
Record Dates: First submitted 2007-09-20; First posted 2007-09-26 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — epinastine; Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Elestat (Experimental)
  Interventions: Drug: Elestat
- Pataday (Active Comparator)
  Interventions: Drug: Pataday

INTERVENTIONS:
Drug: Elestat — Elestat BID for 2 days
  Arms: Elestat
Drug: Pataday — Pataday QD for 2 days
  Arms: Pataday

SUMMARY:
The purpose of this study is to compare the effects of two marked ocular anti-allergy medications in cat sensitive subjects with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of ocular allergy to cats.
* Positive skin prick allergen reaction to cat dander.

Exclusion Criteria:

* Use of any topical or systemic corticosteroids, immunosuppressive agents, antihistamines, decongestants, NSAIDs, or asprin during the two weeks prior to enrollment into the study.
* History of severe asthma, reactive airway disease or bronchial obstruction.
* Ocular surgery or trauma in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Raizman, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Elestat: 1 drop each eye for 2 days
- Pataday: 1 drop each eye for 1 day
Period: Overall Study
Arm/Group | Elestat | Pataday
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elestat | Pataday | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.18) | 40.1 (13.41) | 40.7 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 47
  Male | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Itch Score From Baseline
Description: Ocular itch was measured on a 0 (none) to 4 (severe itch with continual desire to rub eyes) scale. Negative values for change from baseline represent favorable outcomes.
Time Frame: 0 hours, 12 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elestat | Pataday
Number analyzed (Participants) | 40 | 39
units on a scale | -1.5 (1.36) | -1.5 (1.07)
Statistical Analysis 1: Comparison: Elestat vs Pataday; ITT (Intent to Treat); Test type: Superiority or Other; p = 0.532, ANCOVA

2. Secondary Outcome: Ocular Comfort Score at 12 Hours
Description: Ocular comfort was measured on a 0 (more uncomfortable) to 10 (more comfortable) scale.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elestat | Pataday
Number analyzed (Participants) | 40 | 39
units on a scale | 8.6 (1.62) | 8.5 (1.94)
Statistical Analysis 1: Comparison: Elestat vs Pataday; ITT (Intent to Treat); Test type: Superiority or Other; p = 0.927, Student's t-test

ADVERSE EVENTS:
Arm/Group | Elestat | Pataday
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish or discuss trial results until written communication is received from Inspire.